CLINICAL TRIAL: NCT03217539
Title: The Two-County Swedish Mammography Screening Trial
Brief Title: The Swedish Two-County Trial of Mammography Screening
Acronym: WE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Laszlo Tabar, MD, FACR (Hon), Emeritus Professor, Dalarna County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DalarnaCC
Record Dates: First submitted 2017-07-11; First posted 2017-07-14 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Study Population (Experimental): In the experimental arm, women aged 40-74 who were randomly selected to receive an invitation to undergo imaging with periodic single view mammography screening. This arm is referred to as the Active Study Population (ASP)
  Interventions: Diagnostic Test: Imaging
- Passive Study Population (No Intervention): In the no intervention arm, women aged 40-74 who were randomly selected to not receive an invitation to undergo periodic single view mammography screening received usual care. This arm is referred to as the Passive Study Population (PSP)

INTERVENTIONS:
Diagnostic Test: Imaging
  Other Names: Screening mammography
  Arms: Active Study Population

SUMMARY:
Population-based randomized controlled trial carried out in two Swedish counties, Dalarna and Ostergotland to find out the impact of early detection on mortality from breast cancer.

DETAILED DESCRIPTION:
The Swedish Two-county study is a randomized controlled trial of invitation to mammography screening. The trial took place in Kopparberg (W), now called Dalarna, and Ostergotland counties in Sweden. The trial randomized 77,080 women aged 40-74 years to invitation to screening (active study population, ASP) and 55,985 women to no invitation to screening (passive study population, PSP). The trial started in 1977 in W-county and in 1978 in E-county. Women in age 40-49 years were invited to single-view mammography screening on average every 24 months, and women aged 50-74 years on average every 33 months. Approximately seven years after randomization a significant 31% decrease in breast cancer mortality was observed in the ASP group, whereupon the PSP was invited to screening once and the screening phase of the trial ended. The mortality data have been reported every two years during the follow-up period and published in peer-reviewed medical journals. The investigators have follow-up data to the Dec 31 2015. The 29-year follow-up data has been published in 2012 in Radiology. Publication of the long-term data reflects the fact that deaths avoided by early detection include some that would have occurred a considerable time later than the screening.

ELIGIBILITY:
Inclusion criteria

* Female
* Aged 40-74
* No history of breast cancer

Exclusion criteria

• Breast cancer diagnosis prior to randomization

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation
Enrollment: 133065 (Actual)
Dates: Start 1977-07-07 (Actual); Primary Completion 1986-09-09 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Breast cancer death | 9 years
  Comparison of breast cancer mortality in the ASP versus PSP

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo K Tabar, MD, Principal Investigator — Department of Mammography, Falun Central Hospital